CLINICAL TRIAL: NCT06118697
Title: Safety and Feasibility of Aerodigestive Stimulation Therapy in Infants With Complex Feeding Difficulties
Brief Title: Feasibility of Aerodigestive Stimulation Therapy Trial
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sudarshan Jadcherla (Other)
Responsible Party: Sponsor-Investigator, Sudarshan Jadcherla, Principal Investigator, Innovative Feeding Disorders Research Program, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000804
Record Dates: First submitted 2023-10-26; First posted 2023-11-07 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Feeding Disorder Neonatal
Keywords: Chronic tube feeding; Gastrostomy; Deglutition; Esophageal manometry

STUDY DESIGN:
Intervention Model Description: Mechanistic study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants with Complex Feeding Difficulties (Experimental): Weekly manometric esophageal stimulation as well as consistent nutritive oral feeding therapy
  Interventions: Procedure: Esophageal stimulation with high resolution esophageal manometry and nutritive oral feeding therapy

INTERVENTIONS:
Procedure: Esophageal stimulation with high resolution esophageal manometry and nutritive oral feeding therapy — Subjects will be given weekly pharyngo-esophageal stimulation guided by high resolution impedance manometry for 4 weeks. During this time of study intervention, every feed will start with nutritive oral stimulation with at least 5 mL of the infant's prescribed diet.

SUMMARY:
The goal of this study is to demonstrate safety, feasibility, and efficacy of a novel pharyngo-esophageal stimulation technique in restoring aerodigestive and swallowing functions in select infants at-risk for chronic gavage tube feeding or gastrostomy. The main aims are:

* To provide consistent activation of deglutition (the process of swallowing), swallowing-airway interactions, and peristalsis in order to decrease the risk of home tube feeding.
* To examine whether physical and manometric evidence-guided interventions and biofeedback will improve compliance, minimize parental stress, and increase satisfaction and perceived self-confidence with infant feeding.

Participants will have weekly pharyngo-esophageal stimulation guided by High Resolution Impedance Manometry (HRIM) for 4 weeks or until discharge, oral nutritive stimulation of at least 5 mL of prescribed milk with each feed, and weekly parental education and feedback regarding feeding progress.

DETAILED DESCRIPTION:
Stimulation will be provided to the esophagus using esophageal manometry starting at enrollment and then weekly for 4 weeks or until discharge, whichever occurs first. During the 4 weeks of study enrollment, subjects will also be provided nutritive oral feeding therapy with each care with a minimum of 5 mL of their prescribed feed. Feeding evaluations by a study team member will occur once a day during the length of the 4-week trial. The study team will do weekly rounds at the bedside to evaluate feeding progress and study interventions. A feeding plan will be posted at the bedside for clear communication with the care team and family of the subjects.

ELIGIBILITY:
Inclusion Criteria:

* NICU infant ≥37 weeks postmenstrual age not taking full oral feeds
* Consult to Neonatal & Infant Feeding Disorder Program for oral feeding difficulty with diagnostic manometry ordered
* Presence of peristaltic and sphincteric reflexes at initial manometry

Exclusion Criteria:

* Potentially lethal chromosomal anomalies
* Craniofacial malformations
* Foregut malformations

Ages: 1 Day to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Oral feeding volumes prior to and at the completion of the study | Collected at 4 weeks or prior to discharge
  Oral feeding volume will be compared prior to the initial manometry study and after the completion of the final manometry study after 4 weeks or prior to discharge, whichever is earliest
Parent surveys | 4 weeks or prior to discharge
  Parental questionnaires will be compared from prior to initial esophageal manometry study and after completion of final esophageal manometry study.

CONTACTS AND LOCATIONS:
Overall Officials: Sudarshan Jadcherla, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
will revisit at a later date